CLINICAL TRIAL: NCT03806387
Title: Physical and Cognitive Performance During the Two First Years of Lemtrada Treatment - a Prospective Observational Study
Brief Title: Physical and Cognitive Performance During the Two First Years of Lemtrada Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MS_Improve
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab will be given two times, separated by 1 year.
  Other Names: Lemtrada

SUMMARY:
Multiple Sclerosis (MS) is a chronic autoimmune neurodegenerative disease of the central nervous system (CNS). The symptoms of MS are wide-ranging, but patients perceive loss of physical function (gait) and cognitive function as the most critical consequences of the disease. Moreover, recent studies have shown that already at early disease stages functional impairments are present.

One of the more recent approved medical treatments for MS patients is Alemtuzumab (product name Lemtrada), a humanized monoclonal antibody targeting CD52 cells, that depletes and repopulates B lymphocytes and T lymphocytes, causing sustained changes in the adaptive immunity. In 2013 and 2014 Alemtuzumab was approved in EU and USA, respectively.

With the exception of the MS Functional Composite z-score, the previous clinical studies investigating the effect of Alemtuzumab have exclusively focused on clinical parameters such as MRI indications of disease activity (accumulation of lesion, total and regional brain atrophy etc.), relapse-rates, changes in 'expanded disability status scale' (EDSS) and side-effects/adverse events. However, no previous studies have performed in depth monitoring on how physical or cognitive performance are affected following initiation of treatment with Alemtuzumab despite the paramount importance to patients.

The primary purpose of this project is to monitor the changes in physical performance during the first two years of treatment with Alemtuzumab in a well characterised Danish cohort of people with relapsing-remitting MS. A secondary purpose is to monitor the impact of Alemtuzumab treatment on cognition during the first two years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical definite Multiple Sclerosis diagnosis according to the McDonald criteria
* About to commence alemtuzumab (Lemtrada) treatment
* Expanded Disability Status Scale (EDSS) ≤ 5.5
* Signed informed consent

Exclusion Criteria:

* Co-morbidities that prevent participation in the project (dementia, serious cognitive disorders etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis patients will be recruited from MS clinics all over Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Six minute walking test (6MWT) | From baseline to 24 months
  Change in maximal walking distance covered in 6 minutes

SECONDARY OUTCOMES:
Six minute walking test (6MWT) | From baseline to 3 months, 6 months, and 12 months
  Change in maximal walking distance covered in 6 minutes
Timed 25 foot walk (T25FWT) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in maximal walking speed
5 times sit to stand test (5STS) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in time to perform 5 times sit to stand test (5STS)
Timed Up and Go (TUG) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in time to perform Timed Up and Go (TUG)
Stair Climbing test | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in time to perform 9-step stair climbing
Six Spot Step Test (SSST) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in maximal walking speed while challenging coordination/balance
Maximal oxygen uptake (VO2 max) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in aerobic power
Maximal muscle strength | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in isometric and dynamic knee extensor muscle strength, isometric hand grip strength
Neuromuscular activation | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in neural drive during maximal isometric knee extension
Body composition - limb lean mass | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in total lower limb lean mass (kg) (assessed by Dual-energy X-ray Absorptiometry - DXA scan).
Body composition - limb fat mass | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in total lower limb fat mass (kg) (assessed by Dual-energy X-ray Absorptiometry - DXA scan).
Body composition - whole body lean mass | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in total body lean mass (kg) (assessed by Dual-energy X-ray Absorptiometry - DXA scan).
Body composition - whole body fat mass | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in total body fat mass (kg) (assessed by Dual-energy X-ray Absorptiometry - DXA scan).
Selective Reminding Test (SRT) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in cognitive test assessing memory
Symbol Digit Modalities Test (SDMT) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in cognitive test assessing processing speed
Physical activity | From baseline to 3 months, 6 months, 12 months, and 24 months
  Change in accelerometer-based assessment of 24-hour physical activity
Clinical Severity of Disease | From baseline to 3 months, 6 months, 12 months, and 24 months
  Estimation of disease severity by the Expanded Disability Severity Scale (EDSS scores: best 0 = normal neurological exam, worst 10 = death due to multiple sclerosis)
Relapse frequency | From baseline to 3 months, 6 months, 12 months, and 24 months
  Number of relapses
12-item Multiple Sclerosis Walking Scale (MSWS-12) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Self-reported questionnaire assessing impact of MS on walking ability (MSWS-12 scores: best 0, worst 100)
Modified Fatigue Impact Scale (MFIS) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Self-reported questionnaire assessing impact of MS-induced fatigue on a persons life (MFIS total scores: best 0, worst 84; physical subscale scores: best 0, worst 36; cognitive subscale scores: best 0, worst 40; psychosocial subscale scores: best 0, worst 8)
Multiple Sclerosis Impact Scale (MSIS-29) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Self-reported questionnaire assessing impact of MS on day-to-day life, from a physical perspective (MSIS-29 physical scale: best 0, worst 100 (greater impact of disease on daily function = worse health) and from a psychological perspective (MSIS-29 psychological scale: best 0, worst 100 (greater impact of disease on daily function = worse health)
Hospital Anxiety and Depression Scale (HADS) | From baseline to 3 months, 6 months, 12 months, and 24 months
  Self-reported questionnaire assessing impact of MS on anxiety (scores: best 0, worst 21) and depression (scores: best 0, worst 21)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Dalgas, MSc,PhD, Principal Investigator — Aarhus University, Health, Section for Sport Science
Locations (1):
- Aarhus University, Health, Section for Sport Science, Aarhus, Jutland, Denmark

REFERENCES:
- [Derived] Hvid LG, Stenager E, Dalgas U. Objectively assessed physiological, physical, and cognitive function along with patient-reported outcomes during the first 2 years of Alemtuzumab treatment in multiple sclerosis: a prospective observational study. J Neurol. 2022 Sep;269(9):4895-4908. doi: 10.1007/s00415-022-11134-7. Epub 2022 Apr 28. PMID 35482080